CLINICAL TRIAL: NCT04870931
Title: Retrospective Analysis of TEM and TEM-ESD for the Treatment of Rectal Adenomas and Early Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Konstantinos Kouladouros (Other)
Responsible Party: Sponsor-Investigator, Konstantinos Kouladouros, Dr. med. Konstantinos Kouladouros, Universitätsmedizin Mannheim
Organization: Universitätsmedizin Mannheim (Other)
Other Study IDs: UMM01
Record Dates: First submitted 2021-04-28; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Perioperative and Long-term Outcomes of TEM and TEM-ESD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TEM-Group: All patients that underwent TEM
  Interventions: Procedure: TEM / TEM-ESD
- TEM-ESD-Group: All patients that underwent TEM-ESD
  Interventions: Procedure: TEM / TEM-ESD

INTERVENTIONS:
Procedure: TEM / TEM-ESD — Transanal local excision of a rectal tumour as a conventional, full-thickness TEM or submucosal dissection as TEM-ESD

SUMMARY:
We retrospectively analysed all TEM and TEM-ESD procedures that took place in Surgical Clinic of the Municipal Hospital of Karlsruhe and the Surgery Department of the University Hospital of Mannheim from 2007 to 2021. We evaluated the periopüerative and long-term outcomes of both procedures for adenomas, adenocarcinomas and other tumours seperately and we compared the results between the two techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent TEM or TEM-ESD

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We analysed all patients who underwent TEM or TEM-ESD in our centers between 2007 and 2021
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Local recurrence | 5 years

SECONDARY OUTCOMES:
en bloc resection | 5 years
complete en bloc resection | 5 years
procedure time | 5 years
perioperative morbidity | 5 years
long-term adverse events | 5 years
survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Mannheim, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kouladouros K, Baral J. Transanal endoscopic microsurgical submucosal dissection (TEM-ESD) for rectal adenomas: a retrospective cohort study of 145 consecutive cases. Langenbecks Arch Surg. 2022 Sep;407(6):2423-2430. doi: 10.1007/s00423-022-02562-0. Epub 2022 Jun 2. PMID 35652960